CLINICAL TRIAL: NCT05798806
Title: Retrospective, Observational, Multicentric Study Aimed at Developing a Model for Prediction of Axillary Lymph Node Status After Neoadjuvant Chemotherapy in Breast Cancer Patients
Brief Title: Predictive Model of Axillary Nodal Status After Neoadjuvant Chemotherapy in Breast Cancer Patients
Acronym: LNNEO
Status: Active, not recruiting | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Principal Investigator, Fabio Corsi, Professor, Istituti Clinici Scientifici Maugeri SpA
Other Study IDs: 2394
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with diagnosis of cN+ breast cancer who underwent neoadjuvant treatment: Patients with diagnosis of cN+ breast cancer who underwent neoadjuvant treatment and then treated with lymph node biopsy or axillary lymphadenectomy

SUMMARY:
The management of patients diagnosed with breast cancer (BC) with axillary nodal involvement is still a controversial topic. These patients' treatment usually involves the administration of a neoadjuvant chemotherapy (NAC) in order to improve survival rates and increase local disease control. Depending on the tumor subtype, an axillary pathologic complete response (pCR) is achieved in 40-70% of initially axillary node-positive patients (cN+). Concerning patients with an axillary pCR, thus a clinically negative node status (cN0), axillary lymphadenectomy (ALND) might be replaced by less invasive surgical approaches and sentinel lymph node biopsy (SLNB) is considered, in these cases, an effective alternative treatment.

However, the relatively high false negative rates, reported in several validation trials, points out the complexity concerning these patients' treatment. Moreover, histological findings' predictive and prognostic value, after SLNB, of micrometastases and isolated tumor cells (ITCs) is still unclear.

Currently, dual-tracer-guided lymph node biopsy and the surgical removal of ≥ 3 sentinel lymph nodes are known as effective strategies aimed to reduce the false negative rates.

There are several ongoing clinical trials to understand and define the best approach for these patients.

Nowadays, there's great interest in potential prognostic role of systemic inflammation's biochemical markers such as neutrophil-to-lymphocyte ratio (NLR). Systemic inflammation's markers may be nodal pCR's predictors after NAC in node-positive breast cancer patients.

The aim of the study is to develop and validate a pre-operative model, able to predict pCR after NAC to select the patients suitable for a surgery de-escalation strategy.

DETAILED DESCRIPTION:
This is a retrospective, observational, multicentric and no profit study. The study involves patients with diagnosis of cN+ breast cancer who underwent neoadjuvant treatment and then treated with lymph node biopsy or axillary lymphadenectomy, referring to the participating centers.

For each patient the following clinical-anamnestic information will be collected: age, pre-NAC blood cell count, tumor dimension, clinical staging (cT, cN), histological information (tumor subtype, grading, receptors' status, Ki-67 value), neoadjuvant treatment regimen, clinical and radiological local response after NAC, clinical and radiological nodal response after NAC, type of surgery, number of examined lymph nodes, number of positive lymph nodes, pathological staging after surgery (ypT, ypN).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer confirmed by histological examination
* Patients who underwent neoadjuvant chemotherapy
* Axillary lymph nodes involvement at diagnosis (cN≥1), identified by clinical examination and/or imaging techniques and/or axillary lymph node cytology aspirate positive for breast cancer cells.

Exclusion Criteria:

* Patients with M+ at diagnosis
* Contraindications for neoadjuvant chemotherapy

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer is gender based
Study Population: The study involves patients with diagnosis of cN+ breast cancer who underwent neoadjuvant chemotherapy and afterwards treated with lymph node biopsy or axillary lymphadenectomy, referring to the participating centers.
Sampling Method: Probability Sample
Enrollment: 1950 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Selection of features | 48 months
  Identification of pre-operative clinical-pathological features predictive for ypN0 status after NAC in patients with cN+ breast cancer (Logistic regression model will be performed)
Nomogram | 48 months
  Development and validation of a nomogram, based on selected clinical-pathological features, able to predict nodal status after neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri SpA, Pavia, Lombardy, Italy

REFERENCES:
- [Derived] Gasparri ML, Albasini S, Truffi M, Favilla K, Tagliaferri B, Piccotti F, Bossi D, Armatura G, Calcinotto A, Chiappa C, Combi F, Curcio A, Della Valle A, Ferrari G, Folli S, Ghilli M, Listorti C, Mancini S, Marinello P, Mele S, Pertusati A, Roncella M, Rossi L, Rovera F, Segattini S, Sgarella A, Tognali D, Corsi F. Low neutrophil-to-lymphocyte ratio and pan-immune-inflammation-value predict nodal pathologic complete response in 1274 breast cancer patients treated with neoadjuvant chemotherapy: a multicenter analysis. Ther Adv Med Oncol. 2023 Sep 15;15:17588359231193732. doi: 10.1177/17588359231193732. eCollection 2023. PMID 37720495